CLINICAL TRIAL: NCT01148134
Title: Pharmacokinetic Profile of Vincristine Administered Along With Imatinib in the Induction Chemotherapy of Bcr-Abl (Philadelphia Chromosome) Positive Acute Lymphoblastic Leukemia (ALL) Compared to That Without Imatinib in the Treatment of Bcr-Abl Negative ALL Patients
Brief Title: Pharmacokinetic Profile of Vincristine Administered With Imatinib for Bcr-Abl Positive Acute Lymphoblastic Leukemia (ALL) Compared to That Without Imatinib for Bcr-Abl Negative ALL
Status: Terminated | Type: Observational
Why Stopped: Analysis of the first 10 patients did not show anyt trend toward differences in PK profiles between imatinib vs no imatinib groups.
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 10-0300-CE
Record Dates: First submitted 2010-06-18; First posted 2010-06-22 (Estimated); Last update posted 2013-01-11 (Estimated); Status verified 2013-01

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Bcr-Abl positive ALL
- Bcr-Abl negative ALL

SUMMARY:
This study is characterizing the pharmacokinetics of vincristine using two different cohorts of patients. The first cohort includes patients with acute lymphoblastic leukemia (ALL) that are Bcr-Abl positive. This cohort of patients will receive vincristine along with imatinib in the induction chemotherapy regimen. The second cohort includes patients with ALL that are Bcr-Abl negative. This cohort of patients will receive vincristine without imatinib in the induction chemotherapy regimen. This study involves blood draws beginning on day 7 of the treatment protocol and these samples will be analyzed for pharmacokinetic parameters.

Imatinib and vincristine are both metabolized by the hepatic CYP 450 enzyme system. Imatinib is an inhibitor of the system and co-administration of imatinib and vincristine has the potential to increase the blood level of vincristine. This could explain the increased level of neurotoxicity that is currently being seen with the co-administration of these two agents in the treatment of Bcr-Abl positive ALL.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* New Diagnosis of Bcr-Abl positive ALL or Bcr-Abl negative ALL
* Receiving induction chemotherapy with the standard Princess Margaret Hospital modified DFCI protocol
* Will have a functioning central venous access catheter in-situ
* Agreeing to participate in the study and sign the informed consent form

Exclusion Criteria:

* Concomitant use of other agents that inhibit hepatic cytochrome CYP3A4, as these drugs may alter vincristine and imatinib levels
* Elevated liver function tests: bilirubin >1.5xULN or AST/ALT >2.5xULN, or documented history of chronic liver disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Acute Lymphoblastic Leukemia will be selected from the Leukemia Clinic at Princess Margaret Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
To characterize the pharmacokinetics of vincristine in two patient cohorts: Bcr-Abl positive ALL patients treated with the standard protocol with imatinib and Bcr-Abl negative ALL patients treated with the same protocol but without imatinib. | 18-24 months

SECONDARY OUTCOMES:
To determine if there are any objective differences in peripheral neuropathy and ileus between the two groups at Day 14, and to correlate these neurologic assessments with PK results. | 18-24 months

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Brandwein, MD, FRCPC, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada